CLINICAL TRIAL: NCT05891847
Title: Non-interventional Study of Patients With Plexiform Neurofibromas and Neurofibromatosis Type I Starting Selumetinib in Russia
Brief Title: Non-interventional Study of Patients With PN NF1 Starting Selumetinib in Russia
Status: Active, not recruiting | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: D1340R00002
Record Dates: First submitted 2023-03-21; First posted 2023-06-07 (Actual); Last update posted 2025-06-10 (Actual); Status verified 2025-06

CONDITIONS: Neurofibroma
Keywords: NON-INTERVENTIONAL; Selumetinib
MeSH Terms: conditions — Neurofibroma

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Other
Biospecimen Retention: None Retained — n\a, as all procedures will be performed as routine clinical practice
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The purpose of this study is to evaluate the effectiveness, safety of selumetinib and patient's parameters of symptomatic inoperable PN NF1 in real clinical practice in Russia

DETAILED DESCRIPTION:
This study will be non-interventional retrospective and prospective study. Assessment of parameters will be carried out as if a patient is treated in real-life clinical setting. The patients should be enrolled into this project after evaluation of eligibility criteria by an investigator 10 clinical sites. No additional procedures besides those already used in the routine clinical practice will be applied to the patients. Study population will consist of pediatric patients aged 3 years and older with NF1 and symptomatic inoperable PN who were prescribed with selumetinib

ELIGIBILITY:
Inclusion Criteria:

* NF1 diagnosed (according to the criteria for evaluating NF1),
* Symptomatic inoperable PN,
* Patients receiving therapy with selumetinib. For newly treated patients - registration on the first day of starting treatment with selumetinib,
* Age at starting of selumetinib treatment ≥ 3 to ≤ 18 years old (included in the study or started the therapy at the age of 18 years old),
* Patients whose parents or guardians have signed a consent form.

Exclusion Criteria:

* Patients currently participating in an interventional study/clinical trial,
* Patients are excluded if there is evidence of an optic glioma, malignant glioma, malignant peripheral nerve sheath tumor, or other cancer, requiring treatment with chemotherapy or radiation therapy,
* Patients who receive other antitumor treatment options on optic nerve glioma, malignant glioma, malignant tumor of the peripheral nerve sheath, or other cancer. If the patient on selumetinib treatment develop optic nerve glioma, malignant glioma, malignant tumor of the peripheral nerve sheath, or other cancer, he can continue selumetinib therapy +\- other treatment options on physician decision,
* Female patients above 12 age who are pregnant /plan to become pregnant or at breast feeding.

Ages: 3 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Study population will consist of pediatric patients aged 3 years and older with NF1 and symptomatic inoperable PN who were prescribed with selumetinib
Sampling Method: Non-Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2023-03-21 (Actual); Primary Completion 2026-03-20 (Estimated); Study Completion 2026-03-20 (Estimated)

PRIMARY OUTCOMES:
ORR in patients receiving selumetinib according to REiNS criteria | from the FSI date (21 Mar 2023) till 36 months from FSI
  ORR (Overall response rate) in patients receiving selumetinib according to REiNS criteria:
  ORR is defined as the number of patients with CR (complete response) or cPR (confirmed partial response). CR is defined as disappearance of the target lesion. PR is defined as decrease in the volume of the target PN by 20% or more compared to the baseline and is considered unconfirmed at the first detection, confirmed when observed again within 3-6 months, and durable when the response is maintained for 1 year or longer
  In this trial ORR could be taken from the source records of the patient retrospectively. In this case CR or cPR counted from the therapy start date of a patient, which could have been before ICF signing.
Best objective response on selumetinib treatment | from the FSI date (21 Mar 2023) till 36 months from FSI
  a percentage of subjects who achieved a best response of CR, PR or stable disease during treatment
Time to discontinuation of selumetinib | from the FSI date (21 Mar 2023) till 36 months from FSI
Description of diagnostic algorithms for PN NF1 in Russia | from the FSI date (21 Mar 2023) till 36 months from FSI
Reasons for discontinuation of selumetinib | from the FSI date (21 Mar 2023) till 36 months from FSI

SECONDARY OUTCOMES:
Safety: adverse events (date, type, severe grade, seriousness criteria, outcome); | from the FSI date (21 Mar 2023) till 36 months from FSI
Clinical profile of patients with PN NF1 in Russia | from the FSI date (21 Mar 2023) till 36 months from FSI
  features of molecular diagnostics, lesion volume and localization of PN (plexiform neurofibroma)
Demographic profile of patients with PN NF1 in Russia | from the FSI date (21 Mar 2023) till 36 months from FSI
  age, gender of patients
Clinical outcomes of selumetinib treatment | From FSI date (21 Mar 2023) till 36 months from FSI
  changes in PN-associated symptoms

CONTACTS AND LOCATIONS:
Locations (5):
- Russia (5):
  - Research Site, Moscow, Moscow
  - Research Site, Moscow
  - Research Site, Novosibirsk
  - Research Site, Saint Petersburg
  - Research Site, Yekaterinburg